CLINICAL TRIAL: NCT03740490
Title: Smartphone Based Smoking Cessation Intervention
Acronym: Smart-TR01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9860; R01CA221819 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Smartphone Based Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart-T + NRT (Experimental): Smart-T provides content during the pre-quit and post-quit periods to prepare and support participants during their quit attempt. The Smart-T app contains multiple components including an EMA delivery and data transfer system, automated messages based upon EMA responses, and on-demand content. All participants will receive free nicotine replacement therapy (NRT).
  Interventions: Combination Product: Smart-T + NRT
- NCI QuitGuide + NRT (Active Comparator): The National Cancer Institute's QuitGuide app is a free smartphone app and is one of few apps that includes many of the recommendations detailed in the Clinical Practice Guideline. The QuitGuide app aims to help smokers understand their smoking patterns and develop the skills needed to quit smoking. QuitGuide provides content during the pre-quit and post-quit periods to prepare and support participants during their quit attempt. All participants will receive free nicotine replacement therapy (NRT).
  Interventions: Combination Product: QuitGuide + NRT

INTERVENTIONS:
Combination Product: Smart-T + NRT — Smart-Treatment App and Nicotine Replacement Therapy
  Arms: Smart-T + NRT
Combination Product: QuitGuide + NRT — NCI QuitGuide Treatment App and Nicotine Replacement Therapy
  Arms: NCI QuitGuide + NRT

SUMMARY:
Smoking is becoming increasingly concentrated among individuals with the lowest levels of income, education, and occupational status. In fact, smoking rates in the United States among people living below the poverty line is nearly twice as high as those above the poverty threshold. Highly flexible and low burden technology-based treatment approaches may overcome many of the barriers that have limited the use and effectiveness of traditional smoking cessation treatments among low socioeconomic status (SES) adults. Ecological momentary assessment (EMA), in which mobile devices are used to capture moment-to-moment experiences, allows for the measurement of phenomena in real-time within natural settings. Smartphone-based smoking cessation apps could offer easily accessible, highly tailored, and intensive interventions at a fraction of the cost of traditional smoking cessation counseling. The Smart-T app uses a lapse risk estimator to identify moments of heightened risk for lapse, and the algorithm tailors treatment messages in real-time based upon level of imminent smoking lapse risk and currently present lapse triggers. This study will compare smoking cessation rates for those randomized to the Smart-T app or the NCI QuitGuide app.

DETAILED DESCRIPTION:
Smoking is becoming increasingly concentrated among individuals with the lowest levels of income, education, and occupational status. In fact, smoking rates in the United States among people living below the poverty line is nearly twice as high as those above the poverty threshold. Highly flexible and low burden technology-based treatment approaches may overcome many of the barriers that have limited the use and effectiveness of traditional smoking cessation treatments among low SES adults. Ecological momentary assessment (EMA), in which mobile devices are used to capture moment-to-moment experiences, allows for the measurement of phenomena in real-time within natural settings. Smartphone-based smoking cessation apps could offer easily accessible, highly tailored, and intensive interventions at a fraction of the cost of traditional smoking cessation counseling. The Smart-T app uses a lapse risk estimator to identify moments of heightened risk for lapse, and the algorithm tailors treatment messages in real-time based upon level of imminent smoking lapse risk and currently present lapse triggers.

The study aims are to:

Determine the impact of treatment condition (i.e., Smart-T vs. QuitGuide app; n=225 per group) on biochemically verified smoking abstinence. Hypothesis 1: Participants randomly assigned to Smart-T will have significantly higher rates of biochemically-verified abstinence than those assigned to QuitGuide at 26 weeks post-quit.

Determine the effect of Smart-T treatment messages on key lapse risk factors. Hypothesis 2: Smoking urge, stress, and cigarette availability will decline more and cessation motivation will increase more following tailored messages that target these lapse triggers in real-time (Smart-T condition) compared with similar situations wherein no messages are provided (QuitGuide condition).

EXPERIMENTAL DESIGN:

Participants (N=550) will be recruited through the TSET Health Promotion Research Center (HPRC) Tobacco Treatment Research Program (TTRP) which is directed by Dr. Darla Kendzor (Co-I). Participants will also be recruited through advertisements. Individuals seeking smoking cessation services at the TTRP will be given a verbal description of the study during their first visit, and those interested will be screened for study eligibility. Those who respond to study advertisements will complete a brief RedCap screener online (i.e., OKSmokerstudy.com), and those who qualify for the study will contacted by study staff and scheduled for a screening/baseline visit. Consistent with our previous research with low SES populations, we have limited exclusion criteria so that the sample is as broad and representative of the population as possible. Interested individuals will be included in the study if they: 1) earn a score ≥ 4 on the Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF)56 indicating > 6th grade English literacy level (required to complete EMAs; at least 88% of all individuals screened for our EMA studies have met this inclusion criterion), 2) are willing to quit smoking 7 days after the baseline assessment, 3) are ≥ 18 years of age, 4) have an expired CO level ≥ 7 ppm suggestive of current smoking for those who attend in person baseline visits or substantiate smoking status (e.g., produce a pack of cigarettes) during baseline assessments by sending picture of cigarettes to staff 5) are currently smoking ≥ 5 cigarettes per day, 6) have no contraindications to using NRT, 7) agree to complete EMAs and CO tests on a study provided or personal smartphone, 8) have household income < 200% of the federal poverty guideline,57 and 9) agree to complete the 26 week post-quit follow-up assessment over the phone and via EMA.

Eligible and interested individuals will be randomized to 1 of 2 groups: 1) Smart-T smoking cessation intervention plus NRT, or 2) NCI QuitGuide smoking cessation intervention plus NRT. Stratified randomization will be used to assign participants to groups based upon race, sex, and cigarettes smoked per day. Participants will be followed for 27 weeks and will attend either 1 in-person visit or complete phone-based baseline visits. Participants will be prompted to complete daily EMAs and tests of smoking status using a portable, low-cost, carbon monoxide monitor (Bedfont iCO Smokerlyzer) on 3 days each week. This data will be used to address primary (i.e., biochemically verified 7-day point prevalence abstinence at 26 weeks post-quit) and secondary outcomes (e.g., 30-day point prevalence abstinence, number of days to first lapse, longest period of smoking abstinence). Geographic location data will be captured multiple times per day to link characteristics of the present environment (e.g., proximity to tobacco outlets) with cessation-related outcomes. We have already created software that integrates the iCO sensor into our InsightTM mobile application platform.

Sub-Study Update: A sample(n=30) of American Indian/Alaska Native participants who have completed the 6 month follow-up assessment will be asked to participate in another qualitative interview designed to assess the perceived utility and cultural fit of the Smart-T App.Information gathered from these qualitative interviews will be used to culturally modify and then experimentally test a new, culturally tailored, version of the Smart-T app for AI/AN smokers who want to quit smoking. In addition, this will serve as an incredibly valuable training opportunity for an emerging Native American scientist to learn tobacco cessation, mHealth, and qualitative methods research from an interdisciplinary team of leading experts in the field.

PROPOSED PROCEDURE:

Individuals who provide informed consent and meet the study inclusion criteria will complete the baseline assessment in TTRP clinic space (the TTRP is located in Research Parkway in a building that is adjacent to the PI's office). Participants may alternatively complete the baseline assessment via phone calls with study staff. Following the baseline assessment, participants will be given instruction on how to complete phone-based EMAs and carbon monoxide assessments. All participants, regardless of condition, will be compensated for completing the baseline assessments, phone-based follow-up, and EMAs. In addition, participants will complete expired breath carbon monoxide tests using the portable iCO device 3 days per week (weeks 1-27).

Baseline and follow-up measures will assess demographic and smoking characteristics, multiple constructs that are known to be related to lapse (e.g., depression, stress, affect, social support), and document intervention effects (See Table 3 and Appendix). We will also access participant perceptions of each app feature. The Baseline process will take approximately 60-90 minutes to complete and data will be collected either on laptop/tablet computers using Questionnaire Development System (QDS) software or remotely via RedCap surveys. QDS uses a computer-administered self-interview format (i.e., ACASI), which reduces data entry errors and the need to retain paper copies of raw data. Each item appears on the computer screen while the program simultaneously reads the item (participants touch the screen to select answers only after QDS reads each item). Participants wear headphones so that others do not hear the survey items. Participants from our previous studies in similar populations, including those with no computer experience, have reported few problems using the QDS program. Staff will be available to help participants who may have difficulty. The RedCap surveys have been designed to replicate the QDS version as closely as possible. The 26 week post-quit follow-up assessment, which includes a longer EMA (i.e., 20-30 minutes) and a phone call based interview (i.e., The Treatment Improvement Survey, 10-15 minutes) that will be recorded for qualitative analysis.

Participants who own an Android smartphone (OS version 6.0 or higher) will be encouraged to download and use the study app on their own phone. Those who do not own this type of smartphone and those who do not have a data plan will be loaned a Samsung smartphone (or equivalent) for 27 weeks so that they may complete EMAs. Participants will navigate through the EMA program and enter data simply by touching the screen. The study app (i.e., Smart-T app or EMA only app) includes a "Call Staff" function/button that automatically calls study staff (e.g., if they have problems completing EMAs). The EMA app also includes a "Payment" button which, when pressed, indicates the number of EMAs that have been prompted and completed and the current level of compensation based upon the up-to-the-moment percentage of EMAs completed. Smartphones will automatically collect data when on-demand features are accessed for both the QuitGuide and Smart-T groups (e.g., number of times features are used). Use of personal vs. study provided phones will be examined as a covariate in all analyses.

IMPORTANCE OF KNOWLEDGE REASONABLY EXPECTED TO RESULT FROM THE RESEARCH:

Although many smartphone based smoking cessation apps exist, none have been developed and empirically validated via a randomized controlled trial in socioeconomically disadvantaged populations of smokers who are seeking to quit smoking. This study is the next step in a line of research that aims to develop and disseminate effective and automated treatments for smoking cessation for this underserved and understudied population. Thus, the knowledge that will be gained from this study is important. Furthermore, the Smart-T app will allow us to reach a population that frequently lacks access to traditional intervention programs, due to limited availability, income, and/or transportation, among other barriers. In addition, the proposed smartphone app is highly versatile and may be easily modified for use in other populations or communities. The risks to subjects are minimal, especially considering the protections against risks that will be implemented for this study.

ELIGIBILITY:
Inclusion Criteria:

1. earn a score ≥ 4 on the Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF) indicating > 6th grade English literacy level
2. are willing to quit smoking 7 days after the baseline visit
3. are ≥ 18 years of age
4. have an expired CO level ≥ 8 ppm suggestive of current smoking
5. are currently smoking ≥ 5 cigarettes per day
6. have no contraindications to using nicotine replacement therapy (NRT)
7. agree to complete EMAs and CO tests on a study provided or personal smartphone
8. have household income < 200% of the federal poverty guideline
9. agree to complete the 26 week post-quit follow-up assessment over the phone and via EMA

Exclusion Criteria:

1. cannot read, speak, and understand English
2. are < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Businelle, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center - HPRC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hebert ET, Kendzor DE, Vidrine DJ, Langford JS, Kezbers KM, Montgomery A, Chen M, Frank-Pearce SG, Vesely SK, Chen S, Barrett ZCW, Businelle MS. Just-in-Time Adaptive Intervention for Smoking Cessation in Low-Income Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2526691. doi: 10.1001/jamanetworkopen.2025.26691. PMID 40810943

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
Started | 225 | 229
Completed | 170 | 183
Not Completed | 55 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT | Total
Number analyzed (Participants) | 225 | 229 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.4) | 52.0 (11.0) | 52.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 167 | 333
  Male | 59 | 62 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 3 | 13
  Not Hispanic or Latino | 215 | 226 | 441
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 8 | 22
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 59 | 111
  White | 143 | 146 | 289
  More than one race | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-Verified Smoking Cessation
Description: Biochemically confirmed 7-day point prevalence abstinence using the CO criteria cutoff of ≤ 6 ppm
Time Frame: 27 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
Number analyzed (Participants) | 225 | 229
Participants | 37 | 23

2. Secondary Outcome: Change in Urge to Quit Smoking
Description: Urge was assessed using a single ecological momentary assessment (EMA) question: "I feel the urge to smoke." Participants rated this item on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Change scores were calculated by subtracting the pre-message rating from the post-message rating for each prompt. The possible range for the change score is -4 to +4. Higher scores indicate an increase in urge to smoke (worse outcome).
Time Frame: 27 weeks
Population: Mean difference in smoking urge change score between treatment groups (Smart-T vs. QuitGuide), based on a mixed-effects regression model. Confidence interval reflects the model-estimated difference between groups, not within-group means.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
Number analyzed (Participants) | 216 | 220
Score on a scale | 0.053 (0.243) | 0.017 (0.232)
Statistical Analysis 1: Comparison: Smart-T + NRT vs NCI QuitGuide + NRT; Each outcome was modeled using a mixed-effects regression with the change score as the dependent variable and treatment group (Smart-T vs. QuitGuide) as the predictor, restricted to participants who received or would have received that type of message; Test type: Superiority; p = 0.284, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.28 to 0.08]

3. Secondary Outcome: Change in Stress
Description: Stress was assessed using a single ecological momentary assessment (EMA) question: "I feel stressed." Participants rated this item on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Change scores were calculated by subtracting the pre-message rating from the post-message rating for each prompt. The possible range for the change score is -4 to +4. Higher scores indicate an increase in stress (worse outcome).
Time Frame: 27 weeks
Population: Mean difference in stress change score between treatment groups (Smart-T vs. QuitGuide), based on a mixed-effects regression model. Confidence interval reflects the model-estimated difference between groups, not within-group means.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
Number analyzed (Participants) | 216 | 220
Score on a scale | -0.005 (0.164) | -0.031 (0.193)
Statistical Analysis 1: Comparison: Smart-T + NRT vs NCI QuitGuide + NRT; Test type: Superiority; p = 0.477, Mixed Models Analysis; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.11 to 0.24]

4. Secondary Outcome: Change in Perceived Cigarette Availability
Description: Perceived cigarette availability was assessed using a single ecological momentary assessment (EMA) question: "Cigarettes are available to me right now." Participants rated this item on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Change scores were calculated by subtracting the pre-message rating from the post-message rating for each prompt. The possible range for the change score is -4 to +4. Higher scores indicate an increase in perceived cigarette availability (worse outcome).
Time Frame: 27 weeks
Population: Mean difference in cigarette availability change score between treatment groups (Smart-T vs. QuitGuide), based on a mixed-effects regression model. Confidence interval reflects the model-estimated difference between groups, not within-group means.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
Number analyzed (Participants) | 216 | 220
Score on a scale | 0.011 (0.181) | -0.010 (0.116)
Statistical Analysis 1: Comparison: Smart-T + NRT vs NCI QuitGuide + NRT; Test type: Superiority; p = 0.456, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.05 to 0.10]

5. Secondary Outcome: Change in Motivation to Quit Smoking
Description: Motivation to quit smoking was assessed using a single ecological momentary assessment (EMA) question: "I want to quit smoking." Participants rated this item on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Change scores were calculated by subtracting the pre-message rating from the post-message rating for each prompt. The possible range for the change score is -4 to +4. Higher scores indicate an increase in motivation to quit smoking (better outcome).
Time Frame: 27 weeks
Population: Mean difference in cessation motivation change score between treatment groups (Smart-T vs. QuitGuide), based on a mixed-effects regression model. Confidence interval reflects the model-estimated difference between groups, not within-group means.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
Number analyzed (Participants) | 216 | 220
Score on a scale | -0.005 (0.139) | -0.002 (0.118)
Statistical Analysis 1: Comparison: Smart-T + NRT vs NCI QuitGuide + NRT; Test type: Superiority; p = 0.215, Mixed Models Analysis; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.56 to 0.13]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 6 months each participant was involved in the study.
Arm/Group | Smart-T + NRT | NCI QuitGuide + NRT
All-Cause Mortality (participants affected / at risk) | 2/225 | 0/229
Serious Adverse Events (participants affected / at risk) | 0/225 | 0/229
Other Adverse Events (participants affected / at risk) | 0/225 | 0/229

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03740490/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03740490/ICF_001.pdf